CLINICAL TRIAL: NCT02509741
Title: Effect of Nutrition and Lifestyles on Obesity and Chronic Disease in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zeng, Director of Health Management Institue, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHPF2012014
Record Dates: First submitted 2015-07-15; First posted 2015-07-28 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: obesity; nutrition; intervention; food replacement; IOT
MeSH Terms: conditions — Obesity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Educational intervention (Experimental): High-protein and low-GI diet education
  Interventions: Behavioral: Education
- Dietary intervention (Experimental): High-protein and low-GI diet plus education
  Interventions: Behavioral: Education; Dietary Supplement: Food replacement
- Internet-of-things (IOT) monitoring intervention (Experimental): Dietary intervention plus IOT monitoring
  Interventions: Behavioral: Education; Dietary Supplement: Food replacement; Behavioral: IOT monitoring
- control (No Intervention): Routine diet recommendation

INTERVENTIONS:
Behavioral: Education
  Arms: Dietary intervention; Educational intervention; Internet-of-things (IOT) monitoring intervention
Dietary Supplement: Food replacement
  Arms: Dietary intervention; Internet-of-things (IOT) monitoring intervention
Behavioral: IOT monitoring
  Arms: Internet-of-things (IOT) monitoring intervention

SUMMARY:
This research is aimed at verifying the effects of diets with high protein and low glycemic index (GI) on weight management among overweight or obese Chinese adult. Additionally, the investigators intend to verify the effects of two new approaches, including food replacement and Internet-of-things (IOT) monitoring on weight control.

ELIGIBILITY:
Inclusion Criteria:

* Health adult, age:18-65，BMI（kg/m2）:27.0-40.0

Exclusion Criteria:

* Patients under regular medical treatment for chronic diseases like diabetes, hypertension, gout and hyperuricemia.
* The patients with chronic renal diseases or other diseases which impose restrictions on the intake of proteins.
* Mental patients.
* People who suffer from secondary obesity caused by endocrine, metabolic disorders or some central nervous system diseases.
* People who are under medical or surgical weight-loss treatments in the past three months.
* People whose weight fluctuations are not less than 5kg in the past two months；
* People with food allergies.
* Men or women who drink regularly over 25g or 15 g daily,respectively.
* Pregnant women and women who prepare to be pregnant.
* Lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite changes of weight, waist circumference and BMI | 3~5 years
  the measure is a composite
Body composition change is measured by means of Bioelectrical Impedance Analysis (BIA) and CT scan | 3~5 years
Dropout ratio during weight-loss period and maintenance period | 3~5 years

SECONDARY OUTCOMES:
Composite changes in cardiovascular health indicators such as blood pressure, blood glucose, and blood lipids | 3~5 years
Composite changes in inflammatory markers, diet and physical activity level, Leptin and adiponectin, compliance of weight-loss and other indicators | 3~5 years
Composite changes in diet-related behaviors such as satiety, food preferences, social support, appetite, healthy lifestyle and psychological aspects | 3~5 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zeng, MD, Principal Investigator — Chinese PLA General Hospital
Locations (2):
- China (2):
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Hangzhou PLA sanatorium, Hangzhou, Zhejiang